CLINICAL TRIAL: NCT02416908
Title: An Investigator Sponsored Phase I/II Study of CLAG + Selinexor in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study of CLAG + Selinexor in Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201505084
Record Dates: First submitted 2015-03-30; First posted 2015-04-15 (Estimated); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; Cladribine; Granulocyte Colony-Stimulating Factor; plerixafor; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Schedule A (selinexor) (Experimental): * Selinexor will be dosed on Days 1, 5, 10, and 12 of the 28-day cycle. All doses will be 60 mg each PO.
  * Single agent selinexor maintenance may be given at 60 mg on Days 1, 8, 15, and 22 (4 doses per 28 day cycle).
  * Cladribine will be given 5 mg/m^2/day IV once daily on Days 4-8.
  * G-CSF will be given 300 mcg SC once daily on Days 3-8.
  * Cytarabine will be given 2000 mg/m^2/day IV once daily on Days 4-8.
  * Bone marrow biopsy will be performed at baseline, Day 3, at time of hematopoietic recovery, and as clinically indicated to assess treatment response.
  Interventions: Drug: Selinexor; Drug: Cladribine; Drug: G-CSF; Drug: Cytarabine; Procedure: Bone marrow biopsy
- Phase I Schedule B (selinexor) (Experimental): * Selinexor will be dosed on Days 1, 5, 10, 12, 17, and 19 of the 28-day cycle. All doses will be 60 mg each PO.
  * Single agent selinexor maintenance may be given at 60 mg on Days 1, 8, 15, and 22 (4 doses per 28 day cycle).
  * Cladribine will be given 5 mg/m^2/day IV once daily on Days 4-8.
  * G-CSF will be given 300 mcg SC once daily on Days 3-8.
  * Cytarabine will be given 2000 mg/m^2/day IV once daily on Days 4-8.
  * Bone marrow biopsy will be performed at baseline, Day 3, at time of hematopoietic recovery, and as clinically indicated to assess treatment response.
  Interventions: Drug: Selinexor; Drug: Cladribine; Drug: G-CSF; Drug: Cytarabine; Procedure: Bone marrow biopsy
- Phase II (selinexor) (Experimental): * Selinexor will be given at the schedule as determined in Phase 1.
  * Single agent selinexor maintenance may be given at 60 mg on Days 1, 8, 15, and 22 (4 doses per 28 day cycle).
  * Cladribine will be given 5 mg/m^2/day IV once daily on Days 4-8.
  * G-CSF will be given 300 mcg SC once daily on Days 3-8.
  * Cytarabine will be given 2000 mg/m^2/day IV once daily on Days 4-8.
  * Bone marrow biopsy will be performed at baseline, Day 3, at time of hematopoietic recovery, and as clinically indicated to assess treatment response.
  Interventions: Drug: Selinexor; Drug: Cladribine; Drug: G-CSF; Drug: Cytarabine; Procedure: Bone marrow biopsy

INTERVENTIONS:
Drug: Selinexor
  Other Names: KPT-330
Drug: Cladribine
  Other Names: Leustatin®; 2-CdA; 2-Chloro-2'-deoxyadenosine; CdA; Chlorodeoxyadenosine
Drug: G-CSF
  Other Names: Plerixafor; Mozobil®
Drug: Cytarabine
  Other Names: Cytosar-U ®; 1-β-Arabinofuranosylcytosine; Cytosine arabinoside; Ara-C
Procedure: Bone marrow biopsy
  Other Names: Bone marrow aspirate

SUMMARY:
Selinexor has shown single-agent activity in a current phase I study enrolling patients with relapsed/refractory AML with durable complete remissions (CR), complete remissions with incomplete hematologic recovery (CRi), partial remissions (PR), and stable disease (SD) observed. Furthermore, common toxicities included nausea, fatigue, and anorexia and were manageable with supportive care agents. Additionally, CLAG chemotherapy has proven activity in relapsed and refractory AML, and has been shown to be a relatively well tolerated regimen without significant non-hematologic toxicity. Given the established role of CLAG chemotherapy, the single agent activity of selinexor, and their non-overlapping toxicities, the investigators propose a phase I/II open label study of selinexor in combination with CLAG for the treatment of patients with relapsed/refractory AML.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed AML (defined using WHO criteria) with one of the following:

  * Primary refractory disease following ≤ 2 cycles of induction chemotherapy, or
  * First relapse with no prior unsuccessful salvage chemotherapy, or
  * Relapsed or refractory to hypomethylating agent, defined as a lack of response, disease progression, loss of response, or intolerance as deemed by the study investigator
* Age between 18 and 70 years old.
* ECOG performance status ≤ 3
* Adequate organ function as defined below:

  * AST(SGOT), ALT(SGPT), total bilirubin ≤ 2 x IULN except when in the opinion of treating physician is due to direct involvement of leukemia (eg. hepatic infiltration or biliary obstruction due to leukemia) or Gilbert's disease
  * Creatinine clearance >50 ml/min, calculated using the formula of Cockroft and Gault: (140-Age) x Mass (kg) / (72 x Creatinine mg/dL); multiply by 0.85 if female.
  * Left ventricular ejection fraction of ≥ 40% by MUGA scan or echocardiogram
* To ensure that no patient will receive a dose of selinexor >70mg/m^2, body surface area (BSA) calculated by Dubois method must be >1.43 m^2
* Patients should not become pregnant or father a baby while on this study because the drugs in this study can affect an unborn baby. Women should not breastfeed a baby while on this study. It is important patients understand the need to use birth control while on this study. It is not anticipated that female patients enrolling in this study will be able to conceive. However, in the rare event that this is possible, female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Acute promyelocytic leukemia (AML with t(15;17)(q22;q11) and variants).
* Previous treatment with CLAG or other chemotherapy regimen containing both cladribine and cytarabine.
* Colony stimulating factors within 2 weeks of study.
* Active graft versus host disease (GVHD) after allogeneic stem cell transplantation. At least 2 months must have elapsed since completion of an allogeneic stem cell transplantation.
* Less than 2 weeks from the completion of any previous cytotoxic chemotherapy (with the exception of hydroxyurea).
* Concurrent active malignancy under treatment except prostate or breast cancer undergoing treatment with hormonal therapy.
* Treatment with any investigational agent within three weeks prior to first dose in this study.
* Active CNS involvement with leukemia.
* Unstable cardiovascular function:

  * symptomatic ischemia, or
  * uncontrolled clinically significant conduction abnormalities (i.e. ventricular tachycardia on antiarrhythmics are excluded and 1st degree AV block or asymptomatic LAFB/RBBB will not be excluded), or
  * congestive heart failure (CHF) of NYHA class ≥3, or
  * myocardial infarction (MI) within 3 months
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to KPT-330 or other agents used in the study.
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable.
* Any medical condition which, in the investigator's opinion, could compromise the patient's safety.
* Pregnant and/or breastfeeding. Patient must have a negative urine pregnancy test within 5 days of study entry.
* Unable to swallow tablets, or diagnosed malabsorption syndrome, or any other disease significantly affecting gastrointestinal function.
* Known active hepatitis B virus (HBV) or C virus (HCV) infection; or known to be positive for HCV ribonucleic acid (RNA) or HBsAg (HBV surface antigen).
* Known human immunodeficiency virus (HIV) infection.
* Serious psychiatric or medical conditions that could interfere with treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Uy, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened to allow participant enrollment on 06/16/2015 and the study was closed to participant enrollment on 01/22/2018.
Pre-assignment Details: * Principal Investigator decided not to escalate to Schedule B dosing in the interest of generating additional safety data
  * Maintenance Phase patients are patients who were enrolled & treated in Phase I Schedule A or Phase II but met certain criteria to receive maintenance selinexor. Their data will only be included in adverse event results.
Groups:
- Selinexor Maintenance Phase (Optional): * These patients were enrolled and treated in the Phase I Schedule A Arm or the Phase II Arm and if they met the requirements below then they were able to receive maintenance selinexor
  * Available for patients who have achieved a CR or CRi based on post-treatment bone marrow assessment at the time of hematopoietic recovery and are either (1) transplant ineligible or (2) do not have a stem cell transplant donor available
  * 60 mg selinexor on Days 1, 8, 15, and 22 of a 28-day cycle
Period: Dose Escalation Phase
Arm/Group | Phase I Schedule A (Selinexor) | Phase I Schedule B (Selinexor) | Phase II (Selinexor) | Selinexor Maintenance Phase (Optional)
Started | 6 | 0 | 34 | 0
Completed | 6 | 0 | 30 | 0
Not Completed | 0 | 0 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Maintenance Phase
Arm/Group | Phase I Schedule A (Selinexor) | Phase I Schedule B (Selinexor) | Phase II (Selinexor) | Selinexor Maintenance Phase (Optional)
Started | 0 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Although there were no dose-limiting toxicities for the first 6 participants treated according to Schedule A dosing, the Principal Investigator decided not to escalate to Schedule B dosing in the interest of generating additional safety data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Schedule A (Selinexor) | Phase I Schedule B (Selinexor) | Phase II (Selinexor) | Total
Number analyzed (Participants) | 6 | 0 | 34 | 40
Age, Continuous [Median (Full Range); unit: years] | 63.5 [21 to 67] |  | 55 [23 to 70] | 55.5 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 13 | 15
  Male | 4 |  | 21 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0 | 0
  Not Hispanic or Latino | 6 |  | 34 | 40
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 2 | 2
  White | 6 |  | 32 | 38
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 |  | 34 | 40

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Treatment as Measured by Incidence of Grade 3-4 Adverse Events Occurring in >5% of Participants
Description: -All adverse events will be classified using the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Time Frame: From start of treatment until 30 days following last day of study treatment or until the start of a subsequent treatment for AML, whichever came first (41 days)
Population: -Phase I Schedule A Arm and Phase II Arm data was combined as all participants received the same dose and schedule of the study regimen.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Schedule A and Phase II: * Selinexor will be dosed on Days 1, 5, 10, and 12 of the 28-day cycle. All doses will be 60 mg each PO.
  * Cladribine will be given 5 mg/m^2/day IV once daily on Days 4-8.
  * G-CSF will be given 300 mcg SC once daily on Days 3-8.
  * Cytarabine will be given 2000 mg/m^2/day IV once daily on Days 4-8.
  * Bone marrow biopsy will be performed at baseline, Day 3, at time of hematopoietic recovery, and as clinically indicated to assess treatment response.
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
Participants
  Lymphocyte count decreased | 32
  White blood cell decreased | 28
  Hypophosphatemia | 26
  Platelet count decreased | 22
  Neutrophil count decreased | 21
  Hyponatremia | 18
  Anemia | 14
  Hyperglycemia | 11
  Skin infection | 10
  Febrile neutropenia | 8
  Sepsis | 8
  Hypokalemia | 8
  Lung infection | 7
  Alanine aminotransferase increased | 5
  Oral thrush | 4
  Hypoxia | 4
  Hypertension | 4
  Diarrhea | 3
  Nausea | 3
  Edema limbs | 3
  Catheter-related infection | 3
  Hematuria | 3
  Respiratory failure | 3

2. Primary Outcome: Complete Remission Rate (CR + CRi)
Description: * Morphologic complete remission (CR): neutrophil count > 1.0 x 109 /L, platelet count ≥ 100 x 109/L, < 5% bone marrow blasts by morphologic review, no Auer rods, no evidence of extramedullary disease. (No requirements for marrow cellularity, hemoglobin concentration).
  * Morphologic complete remission with incomplete blood count recovery (CRi): same as CR but ANC may be <1000/mcl or platelet count <100,000/mcl
  * Participants in the phase I portion of the study, treated at the MTD will count towards the phase II accrual goal for evaluation of the primary endpoint.
Time Frame: Median follow-up of 34 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
Participants | 18

3. Secondary Outcome: Time to Platelet Engraftment
Description: -Time to platelet engraftment: Defined as the date of the first dose of study drug to the date that the platelet count is >100,000/mm^3 in the absence of platelet transfusions.
Time Frame: 56 days
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
days | 38 [29 to 61]

4. Secondary Outcome: Time to Neutrophil Engraftment
Description: -Time to neutrophil engraftment: Defined as the date of the first dose of study drug to the date that the absolute neutrophil count is >1,000/mm3
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
days | 28 [24 to 58]

5. Secondary Outcome: Event-free Survival
Description: Event-free survival (EFS): Defined as the interval from the date of first dose of study drug to date of treatment failure including progressive disease, recurrence, or discontinuation for any reason (including toxicity, patient preference, initiation of new treatment without documented progression, or death due to any cause).
Time Frame: Up to 2 years (median follow-up of 307 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
months | 6.1 [4.5 to 7.8]

6. Secondary Outcome: Duration of Remission
Description: -Duration of remission (DOR): Defined as the interval from the date complete remission is documented to the date of recurrence.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
months | 9.1 [1.9 to NA] — Upper confidence interval not yet reached.

7. Secondary Outcome: Relapse-free Survival
Description: Relapse-free survival (RFS): For patients achieving a complete remission, defined as the interval from the date of first documentation of a leukemia free state to date of recurrence or death due to any cause.
Time Frame: Median follow-up of 307 days
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 18
days | 152 [6 to 730]

8. Secondary Outcome: Overall Survival
Description: Overall survival (OS): Defined as the date of first dose of study drug to the date of death from any cause. OS will be evaluated at 3 month intervals for at least 12 months and up to a maximum of 2 years.
Time Frame: Up to 2 years (median follow-up of 307 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
months | 7.8 [5.7 to 14.1]

9. Secondary Outcome: Number of Participants Who Were Able to Undergo Hematopoietic Stem Cell Transplantation
Description: Allogeneic stem cell transplant utilization: the number of patients proceeding to allogeneic transplant within 2 months following end of study without any additional salvage therapy following study treatment.
Time Frame: Up to 2 years (median follow-up of 307 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Schedule A and Phase II
Number analyzed (Participants) | 40
Participants | 24

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment until 30 days following last day of study treatment or until the start of a subsequent treatment for AML, whichever comes first.
Description: Although there were no dose-limiting toxicities for the first 6 participants treated according to Schedule A dosing, the Principal Investigator decided not to escalate to Schedule B dosing in the interest of generating additional safety data.
Groups:
- Selinexor Maintenance Phase (Optional): * Available for patients who have achieved a CR or CRi based on post-treatment bone marrow assessment at the time of hematopoietic recovery and are either (1) transplant ineligible or (2) do not have a stem cell transplant donor available
  * 60 mg selinexor on Days 1, 8, 15, and 22 of a 28-day cycle
Arm/Group | Phase I Schedule A (Selinexor) | Phase I Schedule B (Selinexor) | Phase II (Selinexor) | Selinexor Maintenance Phase (Optional)
All-Cause Mortality (participants affected / at risk) | 5/6 | 0/0 | 25/34 | 2/2
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/0 | 14/34 | 1/2
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0 | 34/34 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Schedule A (Selinexor) (N=6) | Phase I Schedule B (Selinexor) (N=0) | Phase II (Selinexor) (N=34) | Selinexor Maintenance Phase (Optional) (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | NA | 0 | 0
Constrictive pericarditis (Cardiac disorders) | 0 | NA | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | NA | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | NA | 1 | 0
Fever (General disorders) | 0 | NA | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | NA | 1 | 0
Bone infection (Infections and infestations) | 1 | NA | 0 | 1
Lung infection (Infections and infestations) | 1 | NA | 1 | 0
Sepsis (Infections and infestations) | 1 | NA | 7 | 0
Sinusitis (Infections and infestations) | 0 | NA | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | NA | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | NA | 1 | 0
Seizure (Nervous system disorders) | 0 | NA | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | 0
Hypotension (Vascular disorders) | 0 | NA | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Schedule A (Selinexor) (N=6) | Phase I Schedule B (Selinexor) (N=0) | Phase II (Selinexor) (N=34) | Selinexor Maintenance Phase (Optional) (N=2)
Anemia (Blood and lymphatic system disorders) | 2 | NA | 14 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | NA | 8 | 0
Atrial fibrillation (Cardiac disorders) | 2 | NA | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | NA | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | NA | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | NA | 0 | 0
Sinus brachycardia (Cardiac disorders) | 0 | NA | 8 | 0
Sinus tachycardia (Cardiac disorders) | 2 | NA | 11 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | NA | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | NA | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | NA | 1 | 0
Blurred vision (Eye disorders) | 1 | NA | 2 | 0
Glaucoma (Eye disorders) | 0 | NA | 1 | 0
Intraretinal hemorrhage (Eye disorders) | 0 | NA | 1 | 0
Photophobia (Eye disorders) | 0 | NA | 1 | 0
Vision changes-acuity (Eye disorders) | 0 | NA | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | NA | 2 | 0
Bloating (Gastrointestinal disorders) | 0 | NA | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | NA | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | NA | 12 | 0
Diarrhea (Gastrointestinal disorders) | 4 | NA | 14 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | NA | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | NA | 1 | 0
Hematemesis (Gastrointestinal disorders) | 0 | NA | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | NA | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | NA | 21 | 0
Nausea (Gastrointestinal disorders) | 5 | NA | 18 | 1
Oral pain (Gastrointestinal disorders) | 0 | NA | 1 | 0
Perirectal fistula (Gastrointestinal disorders) | 0 | NA | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | NA | 1 | 0
Small bowel obstruction (Gastrointestinal disorders) | 1 | NA | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | NA | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | NA | 17 | 1
Chills (General disorders) | 3 | NA | 10 | 0
Edema face (General disorders) | 0 | NA | 1 | 0
Edema limbs (General disorders) | 5 | NA | 16 | 0
Fatigue (General disorders) | 4 | NA | 15 | 0
Fever (General disorders) | 0 | NA | 2 | 0
Hypothermia (General disorders) | 0 | NA | 1 | 0
Infusion related reaction (General disorders) | 1 | NA | 3 | 0
Malaise (General disorders) | 0 | NA | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | NA | 2 | 1
Pain (General disorders) | 0 | NA | 7 | 0
Pain at G-tube insertion site (General disorders) | 0 | NA | 1 | 0
Rigors (General disorders) | 0 | NA | 1 | 0
Hepatic abscess (Hepatobiliary disorders) | 1 | NA | 0 | 0
Bacteremia-Bacillus cereus (Infections and infestations) | 0 | NA | 1 | 0
Bacteremia-Enterococcus faecium/Coagulase negative staphylococcus (Infections and infestations) | 0 | NA | 1 | 0
Bacteremia-Escherichia coli/Enterobacter cloacae (Infections and infestations) | 0 | NA | 1 | 0
Bacteremia-Escherichia coli/pseudomonas aeruginosa (Infections and infestations) | 0 | NA | 1 | 0
Bacteremia-Escherichia coli/streptococcus salvarius (Infections and infestations) | 0 | NA | 1 | 0
Bacteremia-MRSE (Infections and infestations) | 0 | NA | 1 | 0
Bacteremia-Staphylococcus epidermidis (Infections and infestations) | 1 | NA | 1 | 0
Bacteremia-Streptococcus mitis (Infections and infestations) | 0 | NA | 1 | 0
Bacteremia-VRE (Infections and infestations) | 0 | NA | 1 | 0
Bone infection (Infections and infestations) | 0 | NA | 1 | 0
Catheter related infection (Infections and infestations) | 2 | NA | 3 | 0
Clostridium-difficile (Infections and infestations) | 0 | NA | 2 | 0
Endocarditis infective (Infections and infestations) | 0 | NA | 1 | 0
Eye infection (Infections and infestations) | 0 | NA | 1 | 0
Folliculitis (Infections and infestations) | 0 | NA | 1 | 0
Fungemia-Candida parapsilosis disseminated (Infections and infestations) | 0 | NA | 1 | 0
HSV positive lip lesion (Infections and infestations) | 0 | NA | 2 | 0
Infectious hepatic lesions secondary to colitis (Infections and infestations) | 1 | NA | 0 | 0
Lung infection (Infections and infestations) | 1 | NA | 6 | 0
Meningitis (Infections and infestations) | 0 | NA | 1 | 0
Oral thrush (Infections and infestations) | 2 | NA | 4 | 0
Parotitis infectious (Infections and infestations) | 0 | NA | 1 | 0
Sepsis (Infections and infestations) | 1 | NA | 1 | 0
Sinusitis (Infections and infestations) | 0 | NA | 1 | 0
Skin infection (Infections and infestations) | 1 | NA | 10 | 0
Upper respiratory infection (Infections and infestations) | 0 | NA | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | NA | 2 | 0
Bleeding at bone marrow biopsy site (Injury, poisoning and procedural complications) | 0 | NA | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | NA | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | NA | 5 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | NA | 6 | 0
Alanine aminotransferase increased (Investigations) | 6 | NA | 17 | 0
Alkaline phosphatase increased (Investigations) | 3 | NA | 19 | 0
Aspartate aminotransferase increased (Investigations) | 5 | NA | 20 | 1
Blood bilirubin increased (Investigations) | 2 | NA | 17 | 0
Creatinine increased (Investigations) | 0 | NA | 1 | 0
Ejection fraction decreased (Investigations) | 0 | NA | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | NA | 3 | 0
INR increased (Investigations) | 3 | NA | 20 | 0
Lymphocyte count decreased (Investigations) | 5 | NA | 32 | 0
Neutrophil count decreased (Investigations) | 1 | NA | 21 | 2
Platelet count decreased (Investigations) | 3 | NA | 22 | 2
Weight gain (Investigations) | 0 | NA | 1 | 0
Weight loss (Investigations) | 5 | NA | 17 | 0
White blood cell decreased (Investigations) | 3 | NA | 28 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | NA | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | NA | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | NA | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | NA | 11 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | NA | 14 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | NA | 14 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | NA | 6 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | NA | 21 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | NA | 31 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | NA | 5 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | NA | 20 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | NA | 5 | 0
Hyponatremia (Metabolism and nutrition disorders) | 6 | NA | 33 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | NA | 30 | 0
Age indeterminant spinal stress fracture (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | NA | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | NA | 5 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 2 | NA | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | NA | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | NA | 2 | 0
Worsening pain-hip/knees/legs (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | 0
Dizziness (Nervous system disorders) | 1 | NA | 6 | 1
Encephalopathy (Nervous system disorders) | 1 | NA | 1 | 0
Headache (Nervous system disorders) | 2 | NA | 6 | 0
Lethargy (Nervous system disorders) | 1 | NA | 0 | 0
Paresthesia (Nervous system disorders) | 1 | NA | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | NA | 2 | 0
Presyncope (Nervous system disorders) | 0 | NA | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | NA | 1 | 0
Somnolence (Nervous system disorders) | 0 | NA | 6 | 0
Syncope (Nervous system disorders) | 0 | NA | 1 | 0
Altered mental status (Psychiatric disorders) | 0 | NA | 1 | 0
Anxiety (Psychiatric disorders) | 1 | NA | 0 | 0
Confusion (Psychiatric disorders) | 0 | NA | 8 | 0
Delirium (Psychiatric disorders) | 2 | NA | 1 | 0
Depression (Psychiatric disorders) | 1 | NA | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | NA | 2 | 0
Insomnia (Psychiatric disorders) | 1 | NA | 4 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | NA | 5 | 0
Bladder spasm (Renal and urinary disorders) | 0 | NA | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | NA | 13 | 0
Proteinuria (Renal and urinary disorders) | 2 | NA | 18 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | NA | 2 | 0
Urinary urgency (Renal and urinary disorders) | 0 | NA | 1 | 0
Urine output decreased (Renal and urinary disorders) | 0 | NA | 2 | 0
Genital edema (Reproductive system and breast disorders) | 0 | NA | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | NA | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | NA | 4 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 6 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 7 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 5 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | NA | 8 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 2 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | NA | 6 | 0
Lipoma (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | 0
Nasal lesion (Skin and subcutaneous tissue disorders) | 1 | NA | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | NA | 3 | 0
Perianal lesion (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | NA | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | NA | 6 | 0
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | NA | 2 | 0
Sweet's syndrome (Skin and subcutaneous tissue disorders) | 0 | NA | 1 | 0
Hematoma (Vascular disorders) | 1 | NA | 2 | 0
Hypertension (Vascular disorders) | 1 | NA | 4 | 0
Hypotension (Vascular disorders) | 1 | NA | 7 | 0
Phlebitis (Vascular disorders) | 0 | NA | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | NA | 2 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | NA | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT02416908/Prot_SAP_000.pdf